CLINICAL TRIAL: NCT02813148
Title: An Observational Post-Authorization Safety Study (PASS) of MOVENTIG® (Naloxegol) Drug Utilization in Selected European Populations
Brief Title: Naloxegol Drug Utilization Post Authorisation Safety Study
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: D3820R00006
Record Dates: First submitted 2016-06-06; First posted 2016-06-24 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Opioid Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Naloxegol — Non-interventional study of drug utilization

SUMMARY:
This post-authorization observational safety study determines the characteristics of patients prescribed naloxegol at time of first prescription and treatment patterns of naloxegol in follow-up in the United Kingdom (UK), Norway, Sweden, and Germany.

DETAILED DESCRIPTION:
The overall research questions for this study are: 1) What are the demographic, clinical, and treatment characteristics (including dose) at baseline of patients prescribed naloxegol in real-world practice (including the use of naloxegol in non-indicated populations)? and 2) What are the treatment patterns of naloxegol utilization during follow-up?

Primary objectives:

1. To describe the characteristics of patients prescribed naloxegol at time of first prescription (demographics, targeted comorbidities, targeted comedications, provider characteristics, and indication characteristics).
2. To describe any of the following treatment patterns:

   * Discontinuation of naloxegol (permanently during the observation period)
   * Switching from naloxegol to other drug(s) potentially used by patients with opioid induced constipation (OIC)
   * Prescription of other drug(s) potentially used by patients with OIC in the same period when naloxegol is prescribed (augmentation)
   * Restart in the prescription of naloxegol (after temporary discontinuation or treatment holiday)
   * Continuous treatment with naloxegol during the study period
   * Change in dosing

Exploratory objective:

1. To identify predictors of length of naloxegol use

ELIGIBILITY:
Inclusion Criteria:

1. The patient has at least 1 prescription of naloxegol in his/her medical record anytime during the study period.
2. The patient has at least 12 months of computerized records prior to the first prescription of naloxegol (index date)

Exclusion Criteria:

* No exclusion criteria will be applied

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the targeted countries who are newly prescribed naloxegol will be identified for inclusion. Patients analyzed in this study will be those who have at least 12 months of continuous data available prior to first prescription. The number of patients who do not have at least 12 months of prior data will be reported for completeness.
Sampling Method: Non-Probability Sample
Enrollment: 17254 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
discontinuation | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 3 years
  Presence (yes/no) of a patient discontinuing naloxegol (i.e. permanently during the observation period)
Switching | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 3 years
  Presence (yes/no) of a patient switching from naloxegol to other drug(s) potentially used by patients with opioid induced constipation (OIC)
Augmentation | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 3 years
  Presence (yes/no) of a patient augmenting therapy with a prescription of other drug(s) potentially used by patients with OIC in the same period when naloxegol is prescribed
Restart | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 3 years
  Presence (yes/no) of a patient restarting the prescription of naloxegol (after temporary discontinuation or treatment holiday)
Continuous Use | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 3 years
  Presence (yes/no) of a patient continuously treated with naloxegol during the study period
Dose Change | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 3 years
  Presence (yes/no) of a patient changing dosing of naloxegol

CONTACTS AND LOCATIONS:
Overall Officials: Rob Swain, Study Director — Kyowa Kirin, Inc.
Locations (4):
- Research Site, Frankfurt am Main, Germany
- Research Site, Oslo, Norway
- Research Site, Mölndal, Sweden
- Research Site, London, United Kingdom